CLINICAL TRIAL: NCT05589545
Title: Full-arch Rehabilitation of Severely Atrophic Maxillae Through the Use of Polyetheretherketone (PEEK) Prostheses Supported by Zygomatic Implants in Combination With Conventional Implants Through the All-on-4 Concept.
Brief Title: PEEK Prostheses in the All-on-4 Concept Using Zygomatic Implants for Full-arch Rehabilitation.
Acronym: PEEKPilotZyg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Malo Clinic (Other)
Collaborators: Invibio Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEEKPilotZyg
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Prosthesis Survival
Keywords: prosthesis, dental implants, zygomatic implants, PEEK
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Prosthetic full-arch rehabilitation using a PEEK-acrylic resin prosthesis
  Interventions: Device: Prosthetic full-arch rehabilitation using a PEEK-acrylic resin prosthesis

INTERVENTIONS:
Device: Prosthetic full-arch rehabilitation using a PEEK-acrylic resin prosthesis — A prosthetic full-arch rehabilitation of atrophic maxillae using a PEEk-acrylic resin prosthesis supported by an ensemble of standard dental implants and zygomatic dental implants, following the All-on-4 Hybrid Concept.
  Other Names: PEEK prosthesis

SUMMARY:
The goal of this study is to evaluate the outcome of a Poly-ether-ether-ketone - acrylic resin prosthesis for full-arch rehabilitation of the atrophic maxillae through the All-on-4 Hybrid concept (standard and zygomatic implants) after one year of follow-up. The main question it aims to answer is:

- What is the survival outcome of the full-arch implant-supported Poly-ether-ether-ketone - acrylic resin prosthesis? The participants already rehabilitated with dental implants will receive a Poly-ether-ehter-ketone prosthesis as a definitive prosthesis.

DETAILED DESCRIPTION:
Following the previous study on the full-arch rehabilitation of edentulous jaws using hybrid prostheses with polyetheretherketone (PEEK) infrastructure and acrylic resin teeth supported by implants in immediate function inserted through the All-on-4 concept it is necessary to further extend the evaluation to the full-arch rehabilitation of severily atrophic maxillae through the use of the same hybrid prostheses supported by immediate function zygomatic implants inserted alone or in combination with conventional implants. To test this, the study design to be used will be a single-centre, prospective, observational cohort study to evaluate the short term outcome of fixed prosthetic implant-supported rehabilitations. The sample of this study consists in 10 patients consecutively treated. The cohort will be evaluated after 4 to 8 weeks, 6 months, 12 months after connection of the prostheses and annually thereafter as long as the patient is willing, regarding: prosthetic survival, implant survival, marginal bone resorption, incidence of mechanical complications (loosening or fracture of prosthetic components), biological complications (peri-implant infection, suppuration, fistulae, sinus infection, gingival dehiscence), patient tissue reaction, aesthetic examination including staining, color stability and anatomic form; patient assessment of in mouth comfort, overall chewing ability, aesthetics and patient quality of life using the Oral Health Impact Profile OHIP-14 questionnaire; assessment of prosthetic preparation (technician satisfaction) concerning laboratory preparation time, clinical operative time and costs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the Investigator, are able to understand this clinical study, co-operate with the procedures and are willing to return to the clinic for all the required post-operative follow-ups.
* Subjects who are able to give voluntary, written informed consent to participate in this clinical study and from whom consent has been obtained.

Exclusion Criteria:

* Female Subjects who are pregnant.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-ups or treatment outcomes.
* Subjects with any condition that would compromise their participation and follow-up in this clinical study.
* Subjects who are currently enrolled in a clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-07-19 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Survival of the prosthesis | one year
  Evaluation of the survival for the PEEK-acrylic resin implant-supported prosthesis; nominal (survival,failure)

SECONDARY OUTCOMES:
Survival of the implants | one year
  Evaluation of the survival for implants supporting the PEEK-acrylic resin implant-supported prosthesis; nominal (survival,failure)
Incidence of biological complications | one year
  Peri-implant infection, abscess, fistulae, suppuration, sinus infection, gingival dehiscence; Nominal (no incidence, incidence)
Incidence of mechanical complications | one year
  Loosening or fracture of prosthetic components; Nominal (no incidence, incidence)
Marginal bone resorption (standard implants) | one year
  Measured through periapical radiographs, in mm between the implant shoulder and the most apical portion of implant-bone contact; Scale
Patient tissue reaction | one year
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Denture staining | one year
  Veneer staining; 0:heavily stained; 10: no stains
Color stability | one year
  Color stability; 0: heavy discoloration; 10: no discoloration
Anatomic form | one year
  Anatomic form; 0: Complete loss of anatomic form; 10: maintained anatomic form
ln mouth comfort | one year
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Aesthetics | one year
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Overall Chewing ability | one year
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Oral Health Impact Profile | One year
  Oral Health Impact Profile OHIP-14 questionnaire
Laboratory preparation time | one year
  Average laboratory time to produce the finished prosthesis, the active technician time spent in CAD design, Cam mill and veneering.
Clinical operative time | one year
  Average operative time to load the final prosthesis

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A de Araújo Nobre, PhD, Principal Investigator — Director of Research, Development and Education
Locations (1):
- Malo Clinic, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Anonymized database containing the study variables
Supporting Information: SAP
Time Frame: Upon study completion and for 8 years.
Access Criteria: Upon solicitation to the Investigators